CLINICAL TRIAL: NCT06904651
Title: VADIOR: Vantaggi Del Posizionamento Preoperatorio Di Accessi Vascolari Avanzati Ad Inserzione Periferica Nel Paziente DIVA Candidato Ad Intervento Ortopedico
Brief Title: VADIOR: Advantages of Pre-operative Positioning of Peripherally Inserted Vascular Accesses in DIVA Patients Undergoing Orthopedic Surgery
Acronym: VADIOR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Monica La Sala, Medical Doctor - Anaesthesiologist, Istituto Ortopedico Rizzoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PG0003287
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Midline Catheter; Orthopedic Surgery
Keywords: ea-diva score, preoperative positioning of peripheral venous accesses; operating room time save; reduction of operating room cost

STUDY DESIGN:
Intervention Model Description: Prospective observational cost-effectiveness study. A preliminary evaluation of the EA-DIVA score of all patients who are candidates for surgery will be performed; all patients with an EA-DIVA score > or = 8 and referred for pre-operative midline or PICC implantation will be prospectively enrolled; anthropometric, anamnestic and clinical parameters of the patient will be collected; indication for implantation, type and characteristics of the implanted device, site of implantation and implantation times will be established by the members of the Vascular Access Team; the DAV follow-up will be performed every 7 days until discharge and/or removal of the device, recording the appearance of signs or symptoms of infection and/or thrombosis and/or other complications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ALL Patients with EA-DIVA SCORE >8 undergoing all type of orthopedic surgery (Experimental): Pre-operative positioning of advanced peripherally inserted vascular access
  Interventions: Device: pre-operative positioning of peripherally inserted vascular accesses devices such as midline or minimidline

INTERVENTIONS:
Device: pre-operative positioning of peripherally inserted vascular accesses devices such as midline or minimidline — pre-operative positioning of peripherally inserted vascular accesses devices such as midline or minimidline ultrasound guided by dedicated vascular access team

SUMMARY:
Our goal is to demonstrate how a standardized approach that involves the pre-operative implantation of the venous access devices in the DIVA patients (EA-DIVA score> or =8), scheduled for orthopedic surgery, impacts both the intra- and post-operative safety of the patient and the economic savings of our institute. The latter would be achieved both through a reduction in operating room costs and in terms of recovery of operating room hours

DETAILED DESCRIPTION:
Prospective observational cost-effectiveness study. A preliminary evaluation of the EA-DIVA score of all patients who are candidates for surgery will be performed; all patients with an EA-DIVA score > or = 8 and referred for pre-operative midline or PICC implantation will be prospectively enrolled; anthropometric, anamnestic and clinical parameters of the patient will be collected; indication for implantation, type and characteristics of the implanted device, site of implantation and implantation time will be established by the members of the Vascular Access Team; the DAV follow-up will be performed every 7 days until discharge and/or removal of the device, recording the appearance of signs or symptoms of infection and/or thrombosis and/or other complications.

The study setting will be :IRCCS Istituto Ortopedico Rizzoli: all hospitalization departments plus the pre-admission clinic for the enrollment of patients with difficult vascular access, classified according to the EA-DIVA Score; the procedure room of the Post-Operative Intensive Care Unit for the implantation of the devices; hospitalization departments for the post-operative monitoring of any complications

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age (≥ 18 years).
* Patients with a history of documented venous difficulties (DIVA Score > or = 8)
* Candidates for surgery in GA or LRA
* Patients who have signed the informed consent

Exclusion Criteria:

* Patients under 18 years of age
* Patients with medical or anatomical contraindications to DAV placement in the upper limbs

  * Local Contraindications: neuromuscular pathologies (long-standing paresis), osteoarticular (fractures, ankylosis), vascular (presence of active DVT affecting the basilar-subclavian-axillary axis), dermatological (infections, burns), lymphatic (axillary lymphadenectomy)
  * Systemic Contraindications: chronic renal failure grade 3b-4-5, patients on periodic chronic hemodialysis or destined for dialysis, severe thrombocytopenia with platelet count < a 50,000/mm3 (relative contraindication not valid for non-tunneled PICCs, midline and minimidline)
  * Anatomical contraindications: deep veins of the arm of inadequate caliber for the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
OPERATING ROOM TIME SAVING | one year
  Estimate of operating room time savings, calculated as hours/year recovered, otherwise used for intra-operative positioning of such devices and/or emergency invasive devices

CONTACTS AND LOCATIONS:
Overall Officials: Monica La Sala, Medicine- Anaesthesiology, Principal Investigator — IRCCS - Istituto Ortopedico Rizzoli Via di Barbiano 1/10 40136 Bologna Italy
Locations (1):
- IRCCS - Istituto Ortopedico Rizzoli Via di Barbiano 1/10 40136 Bologna Italy, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No